CLINICAL TRIAL: NCT06341894
Title: Efficacy and Safety of Dalpiciclib With Endocrine Therapy as Adjuvant Treatment in Patients With Hormone Receptor-positive, HER2-negative Early Breast Cancer
Brief Title: Efficacy and Safety of Dalpiciclib With Endocrine Therapy as Adjuvant Treatment in HR+/ HER2- Early Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Liu Xiaoan, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBU-II-BC-126
Record Dates: First submitted 2024-02-24; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Dalpiciclib and endocrine therapy
  Interventions: Drug: Dalpiciclib; Drug: Endocrine therapy

INTERVENTIONS:
Drug: Dalpiciclib — CDK4/6 inhibitor dalpiciclib, 100mg orally qd
  Other Names: CDK4/6 inhibitor
Drug: Endocrine therapy — Fulvestrant/AI

SUMMARY:
The investigator conduct a phase II multi-center, open-label trial to evaluate efficacy and safety of dalpiciclib with endocrine therapy as adjuvant treatment in patients with medium /high risk hormone receptor-positive, HER2-negative Early Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years-old
* Patient is female with known menopausal status (postmenopausal or premenopausal/perimenopause)
* Patient with histologically confirmed HR+/HER2- early breast cancer (immunohistochemical ER and/or PR≥10%)
* Histologically confirmed invasive breast cancer with anatomic stages of IIA-IIIC stage (T2-4N0-3M0), of which stage IIA only included T1N1M0
* Patients with or without neoadjuvant or adjuvant chemotherapy/ radiotherapy were eligible for inclusion
* From operation to enrollment should not exceed 12 months
* Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* metastatic disease (Stage IV) or inflammatory breast cancer
* Previous or current history of malignant neoplasms, except for curatively treated:Basal and squamous cell carcinoma of the skin,Carcinoma in situ of the cervix.
* Clinically relevant cardiovascular disease:Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
* A history of allergy to the drugs in this study；
* Unable or unwilling to swallow tablets
* History of gastrointestinal disease with diarrhea as the major symptom.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1163 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
invasive Disease-free Survival (iDFS) | From enrollment until time of events up to 3 years
  Invasive disease-free survival time is defined as the time from date of enrollment until the first disease recurrence or death from any cause

SECONDARY OUTCOMES:
Disease-free Survival (DFS) | From enrollment until time of events up to 3 years
  Disease-free survival time is defined as the time from date of enrollment until the first disease recurrence（including carcinoma in situ）or death from any cause.
AEs and SAEs | From the first administration to one months after the last drug administration，up to one month
  Adverse events and Adverse events and serious adverse events according to CACTE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No